CLINICAL TRIAL: NCT03870568
Title: Functional Assessment in Liver Transplantation
Acronym: FrAILT
Status: Terminated | Type: Observational
Why Stopped: study transitioned from LIRB to CIRB
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 015-243
Record Dates: First submitted 2017-03-10; First posted 2019-03-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis; End Stage Liver Disease
Keywords: frailty; liver transplantation; functional status
MeSH Terms: conditions — Fibrosis; End Stage Liver Disease; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to ensure the equity of the liver allocation process, it is important to create objective, scientifically validated markers of frailty in patients with end-stage liver disease that accurately predict patient outcomes. Many measures have been developed to assess this clinical state in elderly patients, but none have been applied to patients with cirrhosis, a population at increased risk for accelerated functional decline. This protocol is designed to learn more about the effects of functional status (also known as "frailty") in liver transplant patients and patient outcomes both before and after liver transplant.

DETAILED DESCRIPTION:
Subjects in this study will be asked questions regarding functional status and ability to do activities at home. Subjects will also be asked to complete several physical tests to assess functional status. For example, subjects will be asked to stand up from a chair several times, balance with their feet together, and walk down a hall as quickly as possible. Subjects will also be asked to perform a hand grip strength test.

Subjects will be assessed at baseline and at every clinic visit in the pre-transplant setting. Subjects will again be assessed at 3, 6, and 12 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Listed for liver transplantation, or are "listable" - i.e, have undergone formal evaluation and been approved for listing if/when patients achieve high enough priority
* Are seen in the outpatient clinic setting

Exclusion Criteria:

* Have severe hepatic encephalopathy at enrollment (defined by the time to complete the Numbers Connection Test (NCT) > 120 seconds, which is the first test that the participants complete upon enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled from Baylor University Medical Center.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Fried Frailty Index measurements in 300 patients with end-stage liver disease awaiting liver transplantation | 5 years
  Fried Frailty is calculated by combining into one score measurements of:
  * Exhaustion: number of days patient felt exhaustion in the past 7 days
  * Physical activity: has the subject performed any weight bearing activity in the past month? (Possible answers: yes or no).
  * Grip strength test using dynamometer: Three measurements reported in kg.
  * Walking speed in a 13-foot (4 meters) walk: Three measurements reported in seconds
    * Unintentional Weight Loss: report if patient has lost 10 lbs or more in the last year.
    * Minnesota Leisure Time Physical Activity Questionnaire (MNLTPA) calculated as a value of 1 for males with MNLTPA score less than 383 kcal/week and for females with a score less than 270 kcal/week.
  Range of score is 0 to 5 with 0 being not frail and 5 being most frail
Liver Frailty Index measurements in 300 patients with end-stage liver disease awaiting liver transplantation | 5 years
  The following measurements are used individually to assess liver frailty index:
  Chair stands: The patient stands up from a sitting position without using his/her arms. The time (in seconds) the patient requires to complete the task is reported.
  Balance testing: patients must stand up in side by side, semi tandem and tandem positions for 10 seconds each. If the subject can't hold position for 10 seconds, the number of seconds that the subject kept in position is reported. Scoring range is 1.0 to 7.0 with 1.0 to 3.0 being "robust" and 4.5 to 7.0 being "frail"
Numbers Connection test measurements in 300 patients with end-stage liver disease | 5 years
  Patient connects numbers that are scattered at random on a piece of paper. Reported as time (in seconds) taken to connect the numbers.
Work status | 5 years
  Possible answers: working, retired, on disability, other.
Hospitalizations | 5 years
  Possible answers: yes or no. If yes, report #of nights and reason.
Activities of daily living (ADLs) | At 1 year post transplantation
  Six questions about daily activities Scoring: A response of yes to any of the questions receives a value of 1. the ADL score is measured as the sum of the values of the 6 questions. A score of 0 correlates with "most dependent" and a score of 6 is "most independent."
Instrumental Activities of Daily Living (IADLs) | At 1 year post transplantation
  Eight questions about daily activities:
  Scoring: each question can be answered with a score of 0 or 1. The final iADL score is the sum of all values. The range of the score is 0 to 8 with 0 being most dependent and 8 being "most independent.'
36 Item Short Form Survey Instrument (SF-36) | At 1 year post transplantation
  Patient will complete a 36 question questionnaire about quality of life at 1 year post transplantation.

SECONDARY OUTCOMES:
Correlation between frailty and outcomes both before and after liver transplantation. | 5 years
  The association between the subject's frailty score and their pre and post transplant outcomes will be assessed.

OTHER OUTCOMES:
Change in measurements of fried frailty before and after liver transplantation. | 5 years
  The changes in frailty score pre and post transplant will be evaluated.
Change in measurements of liver frailty before and after liver transplantation. | 5 years
  The changes in frailty score pre and post transplant will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: James Trotter, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States